CLINICAL TRIAL: NCT06719973
Title: An Open Label, Multicenter, Phase 1 Study of the PARP1 Inhibitor M9466 in Combination With Carboplatin and Platinum-based Anticancer Therapy (DDRiver 521)
Brief Title: Phase 1 Study of M9466 Combined With Carboplatin and Platinum-based Anticancer Therapy (DDRiver 521)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated due to decision made not to proceed with the clinical trial DDRiver 521, that has not yet commenced enrolment, for strategic reasons.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS202650_0009; 2024-514921-45-00 (Other: EU CTR)
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumors
Keywords: PARP inhibitor; DNA damage repair inhibitor; etoposide; atezolizumab; SCLC
MeSH Terms: interventions — Carboplatin; Etoposide; atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Module 1 (Dose Finding): M9466 + Carboplatin (Experimental)
  Interventions: Drug: M9466; Drug: Carboplatin
- Module 2 Part A (Dose Reassessment): M9466 + Carboplatin + Etoposide + Atezolizumab (Experimental)
  Interventions: Drug: Etoposide; Drug: Atezolizumab; Drug: M9446; Drug: Carboplatin
- Module 2 Part B (Dose Expansion): M9466 + Carboplatin + Etoposide + Atezolizumab (Experimental)
  Interventions: Drug: Etoposide; Drug: Atezolizumab; Drug: M9446; Drug: Carboplatin

INTERVENTIONS:
Drug: M9466 — Participants will receive an escalating doses of M9466 orally in 21-day cycles until disease progression, intolerable toxicity, death, withdrawal of study or study consent, lost to follow-up, or end of study.
  Other Names: HRS-1167
  Arms: Module 1 (Dose Finding): M9466 + Carboplatin
Drug: Carboplatin — Carboplatin will be administered intravenously on Day 1 of each 21-day cycle.
  Arms: Module 1 (Dose Finding): M9466 + Carboplatin
Drug: Etoposide — Etoposide will be administered intravenously as per standard of care.
  Arms: Module 2 Part A (Dose Reassessment): M9466 + Carboplatin + Etoposide + Atezolizumab; Module 2 Part B (Dose Expansion): M9466 + Carboplatin + Etoposide + Atezolizumab
Drug: Atezolizumab — Atezolizumab will be administered intravenously as per standard of care.
  Arms: Module 2 Part A (Dose Reassessment): M9466 + Carboplatin + Etoposide + Atezolizumab; Module 2 Part B (Dose Expansion): M9466 + Carboplatin + Etoposide + Atezolizumab
Drug: M9446 — M9446 dose will be further investigated in Module 2 Part A of the study.
  Other Names: HRS-1167
  Arms: Module 2 Part A (Dose Reassessment): M9466 + Carboplatin + Etoposide + Atezolizumab
Drug: M9446 — M9446 recommended Dose for Expansion (RDE) will be further investigated in Module 2 Part B of the study.
  Other Names: HRS-1167
  Arms: Module 2 Part B (Dose Expansion): M9466 + Carboplatin + Etoposide + Atezolizumab
Drug: Carboplatin — Carboplatin will be administered intravenously as per standard of care.
  Arms: Module 2 Part A (Dose Reassessment): M9466 + Carboplatin + Etoposide + Atezolizumab; Module 2 Part B (Dose Expansion): M9466 + Carboplatin + Etoposide + Atezolizumab

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamic, and preliminary clinical activity of M9466 in combinations with carboplatin in advanced or metastatic refractory solid tumor and with the standard of care (carboplatin, etoposide, and atezolizumab) in treatment-naïve ES-SCLC. The results will support any investigation of carboplatin-based combination anticancer treatments with M9466 as well as the selection of a RP2D of M9466 in combination with carboplatin, etoposide, and atezolizumab for a subsequent ES-SCLC study.

ELIGIBILITY:
Inclusion Criteria:

* Module 1: Locally advanced or metastatic solid tumors that are refractory to standard therapy or for which no standard therapy is judged appropriate by the Investigator (that is [i.e.] participants who have exhausted all standard of care options according to International Guidelines), which may convey clinical benefit from the combination treatment with M9466 and carboplatin and have not received more than 3 lines of prior anticancer therapy in the advanced/metastatic setting Module 2: Histologically or cytologically confirmed treatment-naïve, de novo, extensive stage small cell lung cancer (ES-SCLC), who have no history of systemic treatment for the disease. Participant must be considered suitable to receive carboplatin, etoposide, and atezolizumab as first-line treatment for ES-SCLC
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) less than or equal to (<=) 1 (ECOG PS 2 eligible if considered related to SCLC tumor load in Module 2)
* Have adequate hematological, hepatic, and renal function as defined in the protocol
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Module 1: Persistence of AEs related to any prior treatments that have not recovered to Grade <= 1 by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0 unless AEs are clinically non-significant and /or stable on supportive therapy in the opinion of the Investigator (for example [e.g.] neuropathy or alopecia)
* Module 2: Participant has a history of malignancy within 3 years before the date of enrollment (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, benign prostate neoplasm/hypertropia, or malignancy that in the opinion of the Investigator, is considered cured with minimal risk of recurrence within 3 years)
* Participants with known brain metastases, except if clinically controlled, which is defined as individuals with CNS tumors that are asymptomatic and who do not require steroids for the treatment of CNS tumors
* Life expectancy of less than (<) 3 months
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05-14 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Module 1 and Module 2: Number of Participants with Treatment-Emergent Adverse Events (TEAEs) and Treatment Related TEAEs | Time from signing Informed Consent Form (ICF) up to 30 days after end of study intervention (approximately assessed up to 24 months)
Module 1 and Module 2: Number of Participants with Dose-limiting Toxicity (DLT) | Day 1 up to Day 21 of Cycle 1 (each cycle is of 21 days)

SECONDARY OUTCOMES:
Module 1 and Module 2: Pharmacokinetic (PK) Plasma Concentration of M9466 | Pre-dose up to 6 hours post-dose on Cycle 1 Day 1; Pre-dose on Cycle 1 Day 4 and Cycle 1 Day 8 (each cycle is of 21 days)
Module 1 and Module 2: Objective Response (OR) According to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) Assessed by Investigator | Time from first treatment of study intervention up to planned assessment at 24 months
Module 1 and Module 2: Duration of Response (DoR) According to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) as Assessed by the Investigator | Time from first treatment of study intervention up to planned assessment at 24 months
Module 1 and Module 2: Progression-free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) as Assessed by Investigator | Time from first treatment of study intervention up to planned assessment at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc.

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS202650_0009
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html